CLINICAL TRIAL: NCT05665166
Title: A Phase I-II Study of Cryopreserved Autologous CD34+ Haematopoietic Stem Cells Transduced Ex Vivo with CD11b Lentiviral Vector Encoding Human IDS Tagged with ApoEII in Patients with Neuronopathic Mucopolysaccharidosis Type II (nMPS II, Hunters Syndrome)
Brief Title: Gene Therapy with Modified Autologous Hematopoietic Stem Cells for Patients with Mucopolysaccharidosis Type II
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: CTI Clinical Trial and Consulting Services (Other); Great Ormond Street Hospital for Children NHS Foundation Trust (Other); Manchester University NHS Foundation Trust (Other Government); LifeArc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R125432; 2021-000400-38 (EudraCT Number)
Record Dates: First submitted 2022-12-07; First posted 2022-12-27 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Mucopolysaccharidosis II
MeSH Terms: conditions — Mucopolysaccharidosis II

STUDY DESIGN:
Intervention Model Description: Phase I-II prospective, single-centre, non-randomised, open label, safety and proof of concept study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Autologous CD34+ HSCs transduced ex vivo with CD11B LV encoding human IDS tagged with ApoEII (Experimental)
  Interventions: Genetic: Autologous CD34+ HSCs transduced ex vivo with CD11B LV encoding human IDS tagged with ApoEII

INTERVENTIONS:
Genetic: Autologous CD34+ HSCs transduced ex vivo with CD11B LV encoding human IDS tagged with ApoEII — Autologous CD34+ haematopoietic stem cells from MPS II patients will be genetically modified ex vivo using CD11b.IDS-ApoEII Lentiviral Vector (LV), a self-inactivating (SIN) LV expressing the human codon-optimized IDS gene tagged with ApoEII and regulated by a human CD11b myeloid-specific promoter. These transduced CD34+ HSCs will then be cryopreserved until the time of infusion back to the patients

SUMMARY:
MPS II is a genetic disorder that affects boys. Boys with MPS II are missing a working enzyme known as iduronate-2-sulfatase (IDS) which is needed to break down long sugar chains in the body. When this enzyme is missing, these sugars build up to excess causing damage, and stop organs such as the brain from working properly. Children with MPS II often have progressive symptoms such as developmental delay and physical problems.

The only approved treatment for MPS II is enzyme replacement therapy. This involves a regular infusion of the missing enzyme into the blood stream. But this treatment only helps some symptoms and cannot help problems in the brain.

This study will be the first in human clinical trial to check whether using a gene therapy in children with MPS II is safe and is able to provide enough enzyme to help with disease symptoms. Gene therapy involves changing the genetic information that makes up a person, by taking a correct version of the gene that is needed to make the working IDS enzyme and putting it back into the body. This means that the body can then make the missing enzyme itself. The good thing with this therapy is that the body should be able to make this enzyme forever.

To make sure the therapy is safe and working patients will be closely followed for 2 years.

DETAILED DESCRIPTION:
Mucopolysaccharidosis type II (MPSII, Hunter Syndrome) is a rare paediatric X-linked lysosomal storage disease caused by a deficiency in iduronate-2-sulphatase (IDS), due to a mutation on the IDS gene. IDS is essential for the breakdown of the sugar glycosaminoglycans (GAGs), in particular, heparan sulphate (HS) and dermatan sulphate (DS). Without this enzyme, these sugars accumulate in cells causing damage.

Currently, enzyme replacement therapy (ERT) is the only clinically approved treatment available for MPSII. However, ERT is a supportive therapy and is intended to alleviate symptoms and improve patient quality of life, rather than addressing the pathogenic mechanisms of the disease. To date, there is no effective disease-modifying treatment.

This study aims to recruit 5 patients with MPS II who satisfy the inclusion and exclusion criteria and provide full consent, between 3 months and 22 months of age at screening. The investigational medicinal product (IMP) will be a cell-based gene therapy that uses genetically modified autologous CD34+ haematopoietic stem cells transduced with a lentiviral vector containing the human IDS gene tagged with ApoEII. Patients will be followed up for a minimum of 2 years after gene therapy.

The therapy works by adding the gene therapy to cells taken from the child's body. The cells are then frozen and tested for safety before being given back to the child. To collect the cells, we will give the child some medicine to mobilize hematopoietic stem cells (HSC) from their bone marrow into the blood which can then be easily collected. A working copy of the IDS gene is then placed into these cells in the laboratory (ex vivo). The modified HSCs are then given back to the child via a blood infusion where they can travel to and live in the bone marrow. In the bone marrow compartment, these cells will produce new blood cells that can make the IDS enzyme and can carry it around the whole body, including to the brain. This means the excess sugar chains can be broken down which may help cells to function normally. We think this will reduce MPS II symptoms and may help to prevent damage to the brain.

To make sure the therapy is safe patients will be closely followed for 2 years within this trial. Additional follow up for a minimum 15 years post therapy or as per current guidance will then be offered.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent from a legally authorized guardian.
2. Male, age at consent ≥3 months and ≤22 months.
3. Normal cognitive function or mild cognitive dysfunction (patient has a Development Quotient (DQ) score ≥70 at screening as determined by the Bayley Scale of Infant Development-third edition (BSID-III), cognitive domain), or assessed as normal or only mildly impaired by experienced neuropsychologist.
4. Close male relative with known severe (progressive neuronopathic) phenotype of MPSII, or genotype associated with progressive neuronopathic phenotype. This is to be confirmed by the independent expert reviewers.
5. IDS activity ≤10% of the Lower Limit of Normal as measured in leucocytes or plasma, plus either (1) a normal enzyme activity level of at least one other sulfatase (to rule out multiple sulfatase deficiency) as measured in leucocytes, or (2) a documented mutation in the IDS gene.
6. Medically stable and able to accommodate the protocol requirements, including travel without placing an undue burden on the patient/patient's family, as determined by the CI.
7. Patients and their parents/legal guardians must be willing and able to comply with study restrictions and to commit to attend clinic for the required duration during the study and follow-up period as specified in the protocol.

Exclusion Criteria:

1. The patient has previously received stem cell or gene therapy
2. The patient has received modified intravenous ERT or intra-thecal ERT in a trial setting.
3. Patient currently enrolled in another interventional clinical trial
4. The patient has a history of poorly controlled seizures
5. Hemizygous for mutation known to be associated with non-neuropathic phenotype
6. The patient is currently receiving psychotropic or other medications which, in the CI's opinion, would be likely to substantially confound test results
7. The patient has received any investigational medicinal product (including Genistein) within 30 days prior to the Baseline visit or is scheduled to receive any investigational medicinal product during the course of the study
8. Documented Human Immunodeficiency Virus (HIV) infection (positive HIV RNA and/or anti-p24 antibodies)
9. Malignant neoplasia (except local skin cancer) or a documented history of hereditary cancer syndrome. Patients with a prior successfully treated malignancy and a sufficient follow-up to exclude recurrence (based on oncologist opinion) can be included after discussion and approval by the Medical Monitor
10. Myelodysplasia, cytogenetic alterations characteristic of myelodysplastic syndrome and acute myeloid leukaemia, or other serious haematological disorders
11. The patient has a medical condition or extenuating circumstance that, in the opinion of the CI, might compromise the patient's ability to comply with protocol requirements, the patient's well-being or safety, or the interpretability of the patient's clinical data
12. Visual or hearing impairment sufficient to preclude adequate neurodevelopmental testing
13. Severe behavioural disturbances due to reasons other than MPS II and likely to interfere with protocol compliance, as determined by the CI
14. Known sensitivity to Busulfan
15. The receipt of live vaccinations within 30 days prior to treatment start
16. Known sensitivity to DMSO

Ages: 3 Months to 22 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 5 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the tolerability of the IMP in MPS II patients | Up to 24 months post-IMP delivery
  Adverse events will be recorded and graded according to an adapted Paediatric Clinical Toxicity Scale from the National Institute Allergy and Infectious Diseases (NIAID), Autoimmuno-deficiency Syndrome (AIDS) Division
To assess the safety of the IMP in MPS II patients | Up to 24 months post-IMP delivery
  Presence of replication competent virus and integration events in the leukocytes

SECONDARY OUTCOMES:
IDS enzyme activity in total leukocytes | Baseline, 1, 3, 6, 9, 12, 18 and 24 months post-IMP delivery
  Enzyme within or above normal range measured using an IDS enzyme activity assay
Heparan sulphate in plasma | baseline, 1, 3, 6, 9, 12, 18 and 24 months post-IMP delivery
  Heparan sulphate, the substrate for IDS measured within or above normal range
Heparan sulphate in urine | baseline, 1, 3, 6, 9, 12, 18 and 24 months post-IMP delivery
  Heparan sulphate, the substrate for IDS measured within or above normal range
Glycosaminoglycan (GAG) ratio in urine | baseline, 1, 3, 6, 9, 12, 18 and 24 months post-IMP delivery
  GAG ration measured by dimethylmethylene blue [DMB]
IDS enzyme activity in plasma | Baseline, 1, 3, 6, 9, 12, 18 and 24 months post-IMP delivery
  Enzyme within or above normal range measured using an IDS enzyme activity assay
Heparan sulphate in cerebrospinal fluid (CSF) | baseline, 3, 6, 12, and 24 months post-IMP delivery
  Heparan sulphate, the substrate for IDS measured within or above normal range
IDS enzyme activity in CSF | Baseline, 3, 6, 12, and 24 months post-IMP delivery
  Enzyme within or above normal range measured using an IDS enzyme activity assay
VCN in total leukocytes and the bone marrow | baseline and 1, 3, 6, 9, 12, 18 and 24 months post-IMP delivery
  Measured using PCR
Proportion of cells containing the inserted IDS.ApoEII gene in total bone marrow colony forming units (CFUs) | baseline, 1, 6, 12 and 24 month's post-IMP delivery
  CFU assay performed using isolated CD34+ cells and VCN within colonies measured
IDS enzyme activity in the bone marrow | 12 months and at multiple other visits over time
  Enzyme within or above normal range measured using an IDS enzyme activity assay
Cognitive scores (standard scores, age-equivalent scores and development quotient) | baseline, 6, 12, 18 and 24 months post- IMP delivery
  Measured using the Bayley Scales of Infant Development, 3rd Edition (BSID-III) or Kaufman Assessment Battery for Children, 2nd Edition (KABC-II)
Adaptive behaviour (age-equivalent scores) | baseline, 6, 12, 18 and 24 months post-IMP delivery
  Measured using the Vineland Adaptive Behaviour Scales, 3rd Edition (VABS-III)
Quality of life of patient and parents/caregivers | baseline, 6, 12, 18 and 24 months post-IMP delivery
  Measured using questionnaires

OTHER OUTCOMES:
Dermatan sulphate in cerebrospinal fluid (CSF) | Baseline, 3, 6, 12, and 24 months post-IMP delivery
  Dermatan sulphate, the substrate for IDS measured within or above normal range
Dermatan sulphate in plasma | Baseline, 1, 3, 6, 9, 12, 18 and 24 months post-IMP delivery
  Dermatan sulphate, the substrate for IDS measured within or above normal range
Dermatan sulphate in urine | Baseline, 1, 3, 6, 9, 12, 18 and 24 months post-IMP delivery
  Dermatan sulphate, the substrate for IDS measured within or above normal range
IDS enzyme activity in subpopulations (i.e., CD3+, CD15+, CD19+ cells) | baseline, 1, 3, 6, 9, 12, 18 and 24 months post-IMP delivery
  Measured using IDS enzyme activity assay
VCN in blood subpopulations (CD3+, CD15+, CD19+ cells) | baseline, 1, 3, 6, 9, 12, 18 and 24 months post-IMP delivery
  Measured using RT-qPCR
Obstructive sleep apnoea | baseline, 6, 12 and 24 months post-IMP delivery
  Assessed by polysomnography (using the apnoea-hypopnoea index [AHI])
Anti-IDS antibodies in serum and CSF | baseline, 1, 3, 6, 9, 12, 18 and 24 months post-IMP delivery
  measured from baseline
Audiology (hearing) | baseline, 12 and 24 months post-IMP delivery
  Measured using tympanometry and distortion product optoacoustic emission testing
Height and weight | baseline, 1, 3, 6, 9, 12, 18 and 24 months post-IMP delivery
  Measured by standard calibrated stadiometer from the age they can stand independently, prior to this measuring length
Presence of exploratory biomarkers | baseline, 1, 3, 6, 9, 12, 18 and 24 months post-IMP delivery
Cognitive score (GSV) (BSID-III) or Kaufman Assessment Battery for Children, 2nd Edition (KABC-II) | baseline and 6, 12, 18 and 24 months post-IMP delivery
  Measured using the Bayley Scales of Infant Development, 3rd Edition
Adaptive behaviour (GSV) | baseline and 6, 12, 18 and 24 months post-IMP delivery
  Measured using the Vineland Adaptive Behaviour Scales, 3rd Edition (VABS-III)
Rate of fidelity analysis of neurocognitive assessments | baseline, 6, 12, 18 and 24 months post-IMP delivery
  quality of interactions with team
Parental reported observations of child's development | baseline, 6, 12, 18 and 24 months post-IMP delivery
  Using collated comments
Comparison of neurocognitive data with relevant siblings | baseline to 24 months post-IMP delivery
  Collection of DQ, AE and GSV/GSE scores from equivalent siblings

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wynn, Principal Investigator — Manchester Foundation Trust
Locations (1):
- Manchester University Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No